CLINICAL TRIAL: NCT06508684
Title: Current Status and Influencing Factors of Chinese Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma Undergoing Treatment With Bruton's Tyrosine Kinase Inhibitors
Brief Title: Current Status of BTKi Treatment for CLL/SLL in China
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: PICASSO
Record Dates: First submitted 2024-07-14; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: CLL/SLL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BTK inhibitor treated: investigate the current situation of BTK inhibitor treatment for CLL/SLL patients in China and the related influencing factors, including the efficacy and safety, the drug swith between different BTKis，the BTKi based timed limited therapy, etc
  Interventions: Drug: BTK inhibitor

INTERVENTIONS:
Drug: BTK inhibitor — BTKi can refer to Orelabrutinib, Ibrutinib, Zanubrutinib, and Acalabrutinib

SUMMARY:
BTKi has become the standard treatment regimen for CLL/SLL，there is a lack of large-scale real-world studies on the use status and related influencing factors of BTK inhibitors. Therefore, we plan to conduct this multicenter retrospective cross-sectional study to understand the current situation of BTK inhibitor treatment for CLL/SLL patients in China and the related influencing factors, and to explore more suitable treatment patterns based on this.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients with a confirmed diagnosis of CLL/SLL;
* Received BTK inhibitor treatment between February 2023 and February 2024.

Exclusion Criteria:

* Patients with other types of lymphoma;
* Cases deemed unsuitable for inclusion in this study by the investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CLL/SLL Patient who receiving BTKi treatment
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-13 (Actual); Primary Completion 2025-02-12 (Estimated); Study Completion 2025-07-12 (Estimated)

PRIMARY OUTCOMES:
Patient characteristics of those receiving BTKi treatment | up to one year
  Describe the patient characteristics of those receiving BTKi treatment, including age, gender, etc

SECONDARY OUTCOMES:
overall response rate | up to one year
  Assessed according to the iwCLL2018 criteria
Incidence of adverse reactions | up to one year
  Assessed according to the CTCAE 5.0 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Haematology, the First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital, Nanjin, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No